CLINICAL TRIAL: NCT00006172
Title: Light and Negative Ion Treatment for Chronic Depression
Brief Title: Clinical Trials of Two Non-drug Treatments for Chronic Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #3554/R01 MH42931-02; R01MH042931-02 (NIH)
Record Dates: First submitted 2000-08-11; First posted 2000-08-14 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2008-03

CONDITIONS: Mood Disorders; Depressive Disorders; Depression; Chronic Depression
Keywords: Antidepressive Agents; Chronobiology; Chronotherapy; Circadian rhythms; Depressive Disorder; Ions; Light; Lighting; Mood disorders; Phototherapy.
MeSH Terms: conditions — Mood Disorders; Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- bright light box (Active Comparator): 60 min light therapy shortly after awakening
  Interventions: Device: Bright light box
- high-output negative ion generator (Active Comparator): 60 min high-density exposure shortly after awakening
  Interventions: Device: High-output negative ion generator
- low-output negative ion generator (Placebo Comparator): 60 min low-density exposure shortly after awakening
  Interventions: Device: Low-output negative ion generator

INTERVENTIONS:
Device: Bright light box — 60-min light therapy shortly after awakening
  Arms: bright light box
Device: High-output negative ion generator — 60-min high-density ion exposure shortly after awakening
  Arms: high-output negative ion generator
Device: Low-output negative ion generator — 60-min low-density ion exposure shortly after awakening
  Arms: low-output negative ion generator

SUMMARY:
This study investigates the potential efficacy of two nonpharmacologic treatments for nonseasonal depression, bright light exposure or high-density negative air ion exposure. Treatments are self-administered at home by the patient under close clinical supervision.

DETAILED DESCRIPTION:
Bright light exposure and high-density negative ion exposure have been designed to mimic outdoor environmental conditions and are effective in relieving symptoms of seasonal (winter) depression, but their effectiveness in treating chronic depression has not been explored.

Participants in this 10-week study will have an interview, a complete physical exam, and six one-hour appointments for progress evaluations. They will be randomly assigned to either light or high- or low-dose negative ions. Each treatment must be taken consistently for five weeks at the same time every day, after which treatment is temporarily suspended to determine whether symptoms return. Participants will then have the opportunity to try the alternate active treatment to determine which works best for them. On two occasions, participants will provide saliva samples, used to determine the level of melatonin, a hormone that becomes active at night and indicates whether a person's internal circadian clock is "in sync" with the day-night cycle or is early or late. This diagnostic test for melatonin, which is not yet readily available in medical practice, provides our research participants with unique information that can be used to optimize the timing of future treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depression
* Must be able to maintain a regular sleep schedule

Exclusion Criteria:

* Depression restricted to certain seasons of the year
* Presence of other psychiatric disorders
* Current use of psychotropic medication, except for selective serotonin reuptake inhibitors (SSRIs)
* Current use of recreational drugs or supplements that may affect mood
* Current medical illness or medication that may affect response to antidepressant treatment
* Long-distance travel while participating in the program
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2000-04; Primary Completion 2003-07 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Depression scale score | 5 weeks
  change in score relative to baseline

SECONDARY OUTCOMES:
pineal melatonin onset tme | 5 weeks
  change in melatonin onset phase relative to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Terman, Study Director — NYS Psuchiatric Institute
Locations (2):
- United States (2):
  - Department of Psychology, Wesleyan University, Middletown, Connecticut
  - Columbia Presbyterian Medical Center, New York, New York

REFERENCES:
- [Background] Terman M, Terman JS, Ross DC. A controlled trial of timed bright light and negative air ionization for treatment of winter depression. Arch Gen Psychiatry. 1998 Oct;55(10):875-82. doi: 10.1001/archpsyc.55.10.875. PMID 9783557
- [Background] Kripke DF. Light treatment for nonseasonal depression: speed, efficacy, and combined treatment. J Affect Disord. 1998 May;49(2):109-17. doi: 10.1016/s0165-0327(98)00005-6. PMID 9609674
- See also: Click here for a description of environmental therapies — http://www.cet.org/